CLINICAL TRIAL: NCT00087490
Title: Linezolid in the Treatment of Subjects With Complicated Skin and Soft Tissue Infections Proven to be Due to Methicillin-Resistant Staphylococcus Aureus
Brief Title: Skin Structure Infections With Suspected or Proven Methicillin-Resistant Staphylococcus Aureus (MRSA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5951002
Record Dates: First submitted 2004-07-09; First posted 2004-07-13 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-06

CONDITIONS: Skin/Soft Tissue Infections; Methicillin Resistant Staphylococcus Aureus (MRSA)
MeSH Terms: interventions — Linezolid; Vancomycin

INTERVENTIONS:
Drug: linezolid
Drug: vancomycin

SUMMARY:
To determine if linezolid is superior to vancomycin in the treatment of complicated skin and soft tissue infections due to MRSA in adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with signs or symptoms consistent with infection, and if available, laboratory findings consistent with staphylococcal infection (e.g., Gram stain and culture results).
* Signs and symptoms consistent with infection
* Infection suspected to be due to Methicillin Resistant Staphylococcus Aureus

Exclusion Criteria:

* Subjects who were treated with a previous antibiotic (systemic or topical) with MRSA activity (other than linezolid or vancomycin) for more than 24 hours and treatment extended into the 72 hour period prior to the first dose of study drug, unless documented to be a treatment failure (72 hours of treatment and not responding).
* Subjects with uncomplicated skin or superficial skin structure infection such as superficial/simple cellulitis, impetiginous lesion, furuncle, or simple abscess that only need surgical drainage for cure.
* Subjects excluded with necrotizing fasciitis, gas gangrene, osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1077 (Actual)
Dates: Start 2004-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (100):
- United States (56):
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, San Pedro, California
  - Pfizer Investigational Site, Santa Fe Springs, California
  - Pfizer Investigational Site, Sylmar, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Atlantis, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Blue Ridge, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Decatur, Illinois
  - Pfizer Investigational Site, Hines, Illinois
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, North Chicago, Illinois
  - Pfizer Investigational Site, Northlake, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, West Roxbury, Massachusetts
  - Pfizer Investigational Site, East Lansing, Michigan
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Mpls, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Somers Point, New Jersey
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Ducktown, Tennessee
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Forth Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, St. George, Utah
  - Pfizer Investigational Site, Tacoma, Washington
- Argentina (4):
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Loma Hermosa, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Córdoba
- Belgium (3):
  - Pfizer Investigational Site, Charleroi
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Montigny-le-Tilleul
- Brazil (2):
  - Pfizer Investigational Site, São José do Rio Preto, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Chile (2):
  - Pfizer Investigational Site, Providencia, Santiago Metropolitan
  - Pfizer Investigational Site, Santiago
- Colombia (3):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Floridablanca, Santander Department
- Italy (5):
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Udine
  - Pfizer Investigational Site, Varese
- Pfizer Investigational Site, Kuala Lumpur, Malaysia
- Mexico (3):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Portugal (4):
  - Pfizer Investigational Site, Pragal, Almada
  - Pfizer Investigational Site, Amadora
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Smolensk
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- South Africa (4):
  - Pfizer Investigational Site, Kuilsriver, Western Province
  - Pfizer Investigational Site, Johannesburg
  - Pfizer Investigational Site, Parow
  - Pfizer Investigational Site, Pretoria
- Spain (3):
  - Pfizer Investigational Site, Córdoba, Cordoba
  - Pfizer Investigational Site, Girona, Gerona
  - Pfizer Investigational Site, Seville, Sevilla
- United Kingdom (3):
  - Pfizer Investigational Site, Winchester, Hampshire
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Leeds
- Venezuela (4):
  - Pfizer Investigational Site, Ciudad Bolívar, Bolívar
  - Pfizer Investigational Site, Distrito Capital, Miranda
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Maracaibo, Zulia

REFERENCES:
- [Derived] Puzniak LA, Morrow LE, Huang DB, Barreto JN. Impact of weight on treatment efficacy and safety in complicated skin and skin structure infections and nosocomial pneumonia caused by methicillin-resistant Staphylococcus aureus. Clin Ther. 2013 Oct;35(10):1557-70. doi: 10.1016/j.clinthera.2013.08.001. Epub 2013 Sep 3. PMID 24011955
- [Derived] Itani KM, Biswas P, Reisman A, Bhattacharyya H, Baruch AM. Clinical efficacy of oral linezolid compared with intravenous vancomycin for the treatment of methicillin-resistant Staphylococcus aureus-complicated skin and soft tissue infections: a retrospective, propensity score-matched, case-control analysis. Clin Ther. 2012 Aug;34(8):1667-73.e1. doi: 10.1016/j.clinthera.2012.06.018. Epub 2012 Jul 6. PMID 22770644
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951002&StudyName=Skin%20Structure%20Infections%20with%20Suspected%20or%20Proven%20Methicillin-Resistant%20Staphylococcus%20Aureus%20%28MRSA%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Linezolid: Linezolid intravenous infusion or oral tablets every 12 hours (twice daily) at a dose of 600 milligram (mg). Intravenous infusion was administered over a period of 60-90 minutes. Duration of study treatment was 7 to 14 days except in cases of documented methicillin-resistant Staphylococcus aureus (MRSA) bacteremia where it could be extended to 21 days based upon investigator's discretion.
- Vancomycin: Vancomycin intravenous infusion every 12 hours (twice daily) at a dose of 15 mg per kilogram per dose (15 mg/kg/dose) over a period of at minimum 60 minutes for 7 to 14 days except in cases of documented MRSA bacteremia where it could be extended to 21 days based upon investigator's discretion.
Period: Overall Study
Arm/Group | Linezolid | Vancomycin
Started | 544 | 533
Treated | 537 | 515
Completed | 286 | 264
Not Completed | 258 | 269
Not completed — Death | 6 | 4
Not completed — Adverse Event | 3 | 8
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation or (/) Unspecified | 214 | 201
Not completed — Lost to Follow-Up/participant withdrawal | 28 | 36
Not completed — Randomized but not treated | 7 | 18

BASELINE CHARACTERISTICS:
Groups:
- Linezolid: Linezolid intravenous infusion or oral tablets every 12 hours (twice daily) at a dose of 600 mg. Intravenous infusion was administered over a period of 60-90 minutes. Duration of study treatment was 7 to 14 days except in cases of documented MRSA bacteremia where it could be extended to 21 days based upon investigator's discretion.
- Vancomycin: Vancomycin intravenous infusion every 12 hours (twice daily) at a dose of 15 mg/kg/dose over a period of at minimum 60 minutes for 7 to 14 days except in cases of documented MRSA bacteremia where it could be extended to 21 days based upon investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Linezolid | Vancomycin | Total
Number analyzed (Participants) | 537 | 515 | 1052
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (17.6) | 49.4 (17.2) | 49.5 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 200 | 432
  Male | 305 | 315 | 620

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome in Participants With Baseline Methicillin-Resistant Staphylococcus Aureus (MRSA) at End of Study (EOS) for Per-Protocol (PP) Population
Description: Clinical response (CR) was based primarily on global assessment of clinical presentation of participant made by investigator at evaluation time point. At EOS, CR was evaluated as "success" (cure: resolution of clinical signs or (/) symptoms of infection when compared to baseline); "failure": persistence/progression of baseline signs/symptoms of infection after at least 2 days of treatment/development of new clinical findings consistent with active infection; "unknown": extenuating circumstances precluding classification to 1 of above. "Unknown" was excluded from present analysis.
Time Frame: EOS (6 to 28 days after the last dose of study drug)
Population: PP (EOS)set:who received at least 1 dose of drug, with appropriate diagnosis,MRSA as pathogen,satisfied all key inclusion/exclusion criteria, adequate dosing(failure:2 full days of drug, success:4 full days), observed outcome at EOS unless declared failure prior to visit."N"(number of participants analyzed)=participants evaluable for the measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 227 | 209
Percentage of participants
  Success | 84.1 | 79.9
  Failure | 15.9 | 20.1
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; The percent difference was calculated by percentage of participants cured in linezolid arm minus the percentage of participants cured in vancomycin arm along with 2-sided 95 percent (%) confidence interval (CI); Test type: Non-Inferiority or Equivalence — Linezolid was claimed non-inferior to vancomycin if the lower limit of 95% CI for the difference in cure rate is greater than the Food and Drug Administration (FDA) suggested boundary of delta= -0.10; p = 0.249, Chi-squared; Percent Difference = 4.2, 95% CI 2-sided [-3.0 to 11.5]

2. Secondary Outcome: Clinical Outcome in Participants With Baseline MRSA at End of Treatment (EOT) for PP Population
Description: CR evaluated at EOT visit as "success" (cure: resolution of clinical sign/symptoms of infection when compared with baseline; and improvement: 2/more improvement in clinical sign/symptoms of infection when compared with baseline); "failure": persistence/progression of baseline signs/symptoms of infection after at least 2 days of treatment/development of new clinical findings consistent with active infection; "unknown": extenuating circumstances precluding classification to 1 of above. "Unknown": excluded from present analysis.
Time Frame: EOT (within 72 hours of last dose of study drug)
Population: PP (EOT)set:who received at least 1 dose of drug,with appropriate diagnosis,MRSA as pathogen,satisfied all key inclusion/exclusion criteria,adequate dosing(failure:2 full days of drug,success:4 full days),observed outcome at EOT visit unless declared failure prior to visit."N"(number of participants analyzed)=participants evaluable for the measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 239 | 220
Percentage of participants
  Success | 91.6 | 87.7
  Failure | 8.4 | 12.3
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; The percent difference was calculated by percentage of participants cured in linezolid arm minus the percentage of participants cured in vancomycin arm along with 2-sided 95% CI; Test type: Non-Inferiority or Equivalence — Linezolid was claimed non-inferior to vancomycin if the lower limit of 95% CI for the difference in cure rate is greater than the FDA suggested boundary of delta= -0.10; p = 0.168, Chi-squared; Percent Difference = 3.9, 95% CI 2-sided [-1.7 to 9.5]

3. Secondary Outcome: Clinical Outcome in Participants With Baseline MRSA at EOS for Modified-Intent to Treat (mITT) Population
Description: CR was based primarily on global assessment of clinical presentation of participant made by investigator at evaluation time point. At EOS, CR was evaluated as "success" (cure: resolution of clinical signs/symptoms of infection when compared to baseline); "failure": persistence/progression of baseline signs/symptoms of infection after at least 2 days of treatment/development of new clinical findings consistent with active infection; "unknown": extenuating circumstances precluding classification to 1 of above. "Unknown" was excluded from present analysis.
Time Frame: EOS (6 to 28 days after the last dose of study drug)
Population: mITT population included participants who received at least 1 dose of drug with appropriate diagnosis and MRSA as pathogen."N"(number of participants analyzed)= participants evaluable for the measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 276 | 266
Percentage of participants
  Success | 80.8 | 73.7
  Failure | 19.2 | 26.3
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.048, Chi-squared; Percent Difference = 7.1, 95% CI 2-sided [0.1 to 14.2]

4. Secondary Outcome: Clinical Outcome in Participants With Baseline MRSA at EOT for mITT Population
Description: as for outcome 2
Time Frame: EOT (within 72 hours of last dose of study drug)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 284 | 287
Percentage of participants
  Success | 89.4 | 84.7
  Failure | 10.6 | 15.3
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.090, Chi-squared; Percent Difference = 4.8, 95% CI 2-sided [-0.7 to 10.3]

5. Secondary Outcome: Microbiological Outcome in Participants With Baseline MRSA at EOS for PP Population
Description: Microbiological outcome dichotomized to "success" (eradication: absence of baseline isolate (BI) in culture of original infection site (IS); presumed eradication: participant cured and no specimen available for culture; superinfection: clinically failed or improved with new pathogen identified from primary IS other than BI; colonization: isolate was present but not producing infection) and "failure" (persistence: BI present in original IS; presumed persistence: clinically failed and no specimen available for culture; recurrence: presence of isolate at EOS, that was eradicated at EOT).
Time Frame: EOS (6 to 28 days after the last dose of study drug)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 228 | 209
Percentage of participants
  Success | 75.0 | 68.4
  Failure | 25.0 | 31.6
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.127, Chi-squared; Percent Difference = 6.6, 95% CI 2-sided [-1.9 to 15.0]

6. Secondary Outcome: Microbiological Outcome in Participants With Baseline MRSA at EOT for PP Population
Description: Microbiological outcome dichotomized to "success" (eradication: absence of baseline isolate (BI) in culture of original infection site (IS); presumed eradication: participant cured and no specimen available for culture; superinfection: clinically failed or improved with new pathogen identified from primary IS other than BI; colonization: isolate was present but not producing infection) and "failure" (persistence: BI present in original IS; presumed persistence: clinically failed and no specimen available for culture).
Time Frame: EOT (within 72 hours of last dose of study drug)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 239 | 221
Percentage of participants
  Success | 85.4 | 68.8
  Failure | 14.6 | 31.2
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.000, Chi-squared; Percent Difference = 16.6, 95% CI 2-sided [9.0 to 24.2]

7. Secondary Outcome: Microbiological Outcome in Participants With Baseline MRSA at EOS for mITT Population
Description: as for outcome 5
Time Frame: EOS (6 to 28 days after the last dose of study drug)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 279 | 266
Percentage of participants
  Success | 73.5 | 65.8
  Failure | 26.5 | 34.2
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.051, Chi-squared; Percent Difference = 7.7, 95% CI 2-sided [-0.0 to 15.4]

8. Secondary Outcome: Microbiological Outcome in Participants With Baseline MRSA at EOT for mITT Population
Description: as for outcome 6
Time Frame: EOT (within 72 hours of last dose of study drug)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 285 | 289
Percentage of participants
  Success | 84.2 | 69.2
  Failure | 15.8 | 30.8
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.000, Chi-squared; Percent Difference = 15.0, 95% CI 2-sided [8.2 to 21.8]

9. Secondary Outcome: Number of Participants With Clinical Signs and Symptoms at EOT and EOS for PP Population
Description: Participant's clinical evaluation of signs and symptoms were based on global assessment by investigator at specific timepoints. Signs and symptoms of an active skin or soft tissue infection caused by suspected MRSA included purulent discharge, nonpurulent discharge, erythema, swelling, induration, tenderness, pain and local skin warmth. It was recorded by the sponsor using wound parameter score ranging from 0 to 3; "0= none, 1= mild, 2= moderate and 3= severe".
Time Frame: EOT (within 72 hours of last dose of study drug), EOS (6 to 28 days after the last dose of study drug)
Population: PP set:who received at least 1 dose of drug, with appropriate diagnosis,MRSA as pathogen, satisfied all key inclusion/exclusion criteria, adequate dosing(failure:2 full days of drug, success:4 full days),observed outcome at EOS visit unless declared failure prior to the visit.Here,'n'=participants evaluable for specific clinical signs and symptoms.
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 229 | 210
Participants
  Purulent discharge (mild) (EOT) (n=222, 206) | 21 | 17
  Purulent discharge (moderate) (EOT) (n=222, 206) | 1 | 5
  Purulent discharge (severe) (EOT) (n=222, 206) | 0 | 3
  Non-purulent discharge (mild) (EOT) (n=222, 206) | 54 | 57
  Non-purulent discharge (moderate) (EOT)(n=222,206) | 3 | 5
  Non-purulent discharge (severe) (EOT) (n=222, 206) | 0 | 0
  Erythema (mild) (EOT) (n=222, 206) | 53 | 62
  Erythema (moderate) (EOT) (n=222, 206) | 1 | 4
  Erythema (severe) (EOT) (n=222, 206) | 0 | 1
  Swelling (mild) (EOT) (n=222, 205) | 39 | 44
  Swelling (moderate) (EOT) (n=222, 205) | 4 | 6
  Swelling (severe) (EOT) (n=222, 205) | 1 | 1
  Induration (mild) (EOT) (n=222, 206) | 57 | 67
  Induration (moderate) (EOT) (n=222, 206) | 3 | 3
  Induration (severe) (EOT) (n=222, 206) | 0 | 0
  Tenderness (mild) (EOT) (n=222, 206) | 62 | 52
  Tenderness (moderate) (EOT) (n=222, 206) | 4 | 15
  Tenderness (severe) (EOT) (n=222, 206) | 0 | 2
  Pain (mild) (EOT) (n=222, 206) | 38 | 43
  Pain (moderate) (EOT) (n=222, 206) | 4 | 15
  Pain (severe) (EOT) (n=222, 206) | 0 | 2
  Local skin warmth (mild) (EOT) (n=222, 205) | 14 | 19
  Local skin warmth (moderate) (EOT) (n=222, 205) | 0 | 1
  Local skin warmth (severe) (EOT) (n=222, 205) | 0 | 0
  Purulent discharge (mild) (EOS) (n=228, 209) | 10 | 21
  Purulent discharge (moderate) (EOS) (n=228, 209) | 2 | 4
  Purulent discharge (severe) (EOS) (n=228, 209) | 1 | 0
  Non-purulent discharge (mild) (EOS) (n=227, 209) | 35 | 43
  Non-purulent discharge (moderate) (EOS)(n=227,209) | 3 | 2
  Non-purulent discharge (severe) (EOS) (n=227, 209) | 0 | 0
  Erythema (mild) (EOS) (n=228, 209) | 25 | 31
  Erythema (moderate) (EOS) (n=228, 209) | 4 | 6
  Erythema (severe) (EOS) (n=228, 209) | 0 | 0
  Swelling (mild) (EOS) (n=227, 208) | 23 | 25
  Swelling (moderate) (EOS) (n=227, 208) | 0 | 4
  Swelling (severe) (EOS) (n=227, 208) | 1 | 0
  Induration (mild) (EOS) (n=227, 209) | 28 | 37
  Induration (moderate) (EOS) (n=227, 209) | 1 | 1
  Induration (severe) (EOS) (n=227, 209) | 0 | 0
  Tenderness (mild) (EOS) (n=227, 209) | 29 | 32
  Tenderness (moderate) (EOS) (n=227, 209) | 5 | 4
  Tenderness (severe) (EOS) (n=227, 209) | 0 | 0
  Pain (mild) (EOS) (n=227, 209) | 32 | 27
  Pain (moderate) (EOS) (n=227, 209) | 5 | 4
  Pain (severe) (EOS) (n=227, 209) | 0 | 0
  Local skin warmth (mild) (EOS) (n=227, 208) | 11 | 15
  Local skin warmth (moderate) (EOS) (n=227, 208) | 0 | 2
  Local skin warmth (severe) (EOS) (n=227, 208) | 0 | 0

10. Secondary Outcome: Number of Participants With Clinical Signs and Symptoms at EOT and EOS for mITT Population
Description: Participant's clinical evaluation of signs and symptoms were based on global assessment by investigator at specific timepoints. Signs and symptoms of an active skin or soft tissue infection caused by suspected MRSA included purulent discharge, nonpurulent discharge, erythema, swelling, induration, tenderness, pain and local skin warmth. It was recorded using wound parameter score ranging from 0 to 3; "0= none, 1= mild, 2= moderate and 3= severe".
Time Frame: EOT (within 72 hours of last dose of study drug), EOS (6 to 28 days after the last dose of study drug)
Population: mITT population included participants who received at least 1 dose of drug with appropriate diagnosis caused by MRSA. Here, 'n' signified participants who were evaluable and analyzed for specific clinical signs and symptoms.
Measure: Number; unit: Partcipants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 322 | 318
Partcipants
  Purulent discharge (mild) (EOT) (n=286, 292) | 27 | 25
  Purulent discharge (moderate) (EOT) (n=286, 292) | 3 | 9
  Purulent discharge (severe) (EOT) (n=286, 292) | 0 | 3
  Non-purulent discharge (mild) (EOT) (n=286, 292) | 71 | 93
  Non-purulent discharge (moderate) (EOT)(n=286,292) | 5 | 6
  Non-purulent discharge (severe) (EOT) (n=286, 292) | 0 | 0
  Erythema (mild) (EOT) (n=286, 292) | 72 | 88
  Erythema (moderate) (EOT) (n=286, 292) | 3 | 10
  Erythema (severe) (EOT) (n=286, 292) | 1 | 1
  Swelling (mild) (EOT) (n=286, 291) | 54 | 82
  Swelling (moderate) (EOT) (n=286, 291) | 7 | 9
  Swelling (severe) (EOT) (n=286, 291) | 1 | 1
  Induration (mild) (EOT) (n=286, 292) | 73 | 89
  Induration (moderate) (EOT) (n=286, 292) | 6 | 6
  Induration (severe) (EOT) (n=286, 292) | 0 | 0
  Tenderness (mild) (EOT) (n=286, 292) | 77 | 85
  Tenderness (moderate) (EOT) (n=286, 292) | 9 | 22
  Tenderness (severe) (EOT) (n=286, 292) | 1 | 2
  Pain (mild) (EOT) (n=286, 292) | 55 | 194
  Pain (moderate) (EOT) (n=286, 292) | 10 | 20
  Pain (severe) (EOT) (n=286, 292) | 0 | 3
  Local skin warmth (mild) (EOT) (n=286, 290) | 20 | 38
  Local skin warmth (moderate) (EOT) (n=286, 290) | 2 | 3
  Local skin warmth (severe) (EOT) (n=286, 290) | 0 | 0
  Purulent discharge (mild) (EOS) (n=286, 270) | 13 | 28
  Purulent discharge (moderate) (EOS) (n=286, 270) | 4 | 7
  Purulent discharge (severe) (EOS) (n=286, 270) | 1 | 1
  Non-purulent discharge (mild) (EOS) (n=285, 270) | 46 | 56
  Non-purulent discharge (moderate) (EOS)(n=285,270) | 5 | 4
  Non-purulent discharge (severe) (EOS) (n=285, 270) | 0 | 0
  Erythema (mild) (EOS) (n=286, 270) | 40 | 45
  Erythema (moderate) (EOS) (n=286, 270) | 6 | 12
  Erythema (severe) (EOS) (n=286, 270) | 0 | 0
  Swelling (mild) (EOS) (n=285, 269) | 33 | 36
  Swelling (moderate) (EOS) (n=285, 269) | 2 | 11
  Swelling (severe) (EOS) (n=285, 269) | 1 | 1
  Induration (mild) (EOS) (n=285, 270) | 37 | 44
  Induration (moderate) (EOS) (n=285, 270) | 2 | 6
  Induration (severe) (EOS) (n=285, 270) | 0 | 1
  Tenderness (mild) (EOS) (n=284, 270) | 49 | 46
  Tenderness (moderate) (EOS) (n=284, 270) | 6 | 7
  Tenderness (severe) (EOS) (n=284, 270) | 0 | 2
  Pain (mild) (EOS) (n=285, 270) | 49 | 40
  Pain (moderate) (EOS) (n=285, 270) | 7 | 7
  Pain (severe) (EOS) (n=285, 270) | 0 | 3
  Local skin warmth (mild) (EOS) (n=285, 269) | 20 | 27
  Local skin warmth (moderate) (EOS) (n=285, 269) | 0 | 4
  Local skin warmth (severe) (EOS) (n=285, 269) | 0 | 1

11. Secondary Outcome: Duration of Hospital Stay for PP Population
Description: Duration of Hospital Stay was defined as the number of days the participant was cared as an inpatient in the hospital during the maximum 34 days of the study period. The number of days in the hospital was counted from start of study medication to date of discharge or last date known to be in the hospital (for missing discharge dates and participants who died) or Day 34 for participants who continued hospitalization beyond EOS period.
Time Frame: Baseline up to EOS (6 to 28 days after the last dose of study drug)
Population: PP set:who received at least 1 dose of drug,with appropriate diagnosis,MRSA as pathogen,satisfied all key inclusion/exclusion criteria, adequate dosing(failure:2 full days of drug, success:4 full days), observed outcome at EOS visit unless declared failure prior to visit.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 229 | 210
Days | 7.6 (0.44) | 8.9 (0.48)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Null hypothesis was that there was no difference in the length of hospital stay between the treatment groups; Test type: Superiority or Other; p = 0.022, Wilcoxon (Mann-Whitney) — Alpha = 0.05 was the level of significance if the null hypothesis was rejected

12. Secondary Outcome: Duration of Hospital Stay for mITT Population
Description: as for outcome 11
Time Frame: Baseline up to EOS (6 to 28 days after the last dose of study drug)
Population: mITT population included participants who received at least 1 dose of drug with appropriate diagnosis and MRSA as pathogen.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 322 | 318
Days | 7.7 (0.39) | 8.9 (0.40)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Null hypothesis was that there was no difference in the length of hospital stay between the treatment groups; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney) — Alpha = 0.05 was the level of significance if the null hypothesis was rejected

13. Secondary Outcome: Duration of Intravenous Therapy for PP Population
Description: Duration of intravenous antibiotic treatment was measured as the number of days intravenous doses of study medication was administered, before and after discharge.
Time Frame: Baseline up to EOS (6 to 28 days after the last dose of study drug)
Population: PP set:who received at least 1 dose of drug,with appropriate diagnosis,MRSA as pathogen,satisfied all key inclusion/exclusion criteria, adequate dosing(failure:2 full days of drug, success:4 full days), observed outcome at EOS visit unless declared failure prior to visit."N"(number of participants analyzed) = participants evaluable for the measure.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 136 | 210
Days | 5.6 (0.35) | 10.4 (0.22)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Test type: Superiority or Other; p = 0.000, t-test, 2 sided

14. Secondary Outcome: Duration of Intravenous Therapy for mITT Population
Description: as for outcome 13
Time Frame: Baseline up to EOS (6 to 28 days after the last dose of study drug)
Population: mITT population included participants who received at least 1 dose of drug with appropriate diagnosis caused by MRSA. "N"(number of participants analyzed)=participants evaluable for the measure.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 188 | 318
Days | 5.3 (0.28) | 9.8 (0.22)
Statistical Analysis 1: Comparison: Linezolid vs Vancomycin; Test type: Superiority or Other; p = 0.000, t-test, 2 sided

15. Secondary Outcome: Number of Participants Using Medical Resources
Description: Medical resources utilization included a daily log of the participants' location in the hospital and outside of the hospital (non-hospital location), adjusted duration of stay (difference between duration of stay and the duration of discharge delay) and daily log of study drug dosing.
Time Frame: Baseline up to EOS (6 to 28 days after the last dose of study drug)
Population: Data was not analyzed for the primary reporting.
Measure: Number; unit: Participants
Arm/Group | Linezolid | Vancomycin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Linezolid | Vancomycin
Serious Adverse Events (participants affected / at risk) | 31/537 | 32/515
Other Adverse Events (participants affected / at risk) | 250/537 | 250/515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linezolid (N=537) | Vancomycin (N=515)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Brain death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 3
Abscess neck (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Burn infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cellulitis gangrenous (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 0
Intestinal gangrene (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 2
Postoperative wound infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine increased (Investigations) | 0 | 1
Blood culture positive (Investigations) | 1 | 1
Body temperature increased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombectomy (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 0 | 1
Aortic thrombosis (Vascular disorders) | 0 | 1
Arterial rupture (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linezolid (N=537) | Vancomycin (N=515)
Anaemia (Blood and lymphatic system disorders) | 10 | 10
Eosinophilia (Blood and lymphatic system disorders) | 0 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypothrombinaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 3 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Factor XII deficiency (Congenital, familial and genetic disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1
Glaucoma (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 15 | 17
Diarrhoea (Gastrointestinal disorders) | 39 | 14
Dry mouth (Gastrointestinal disorders) | 6 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Faecalith (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Ileal fistula (Gastrointestinal disorders) | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 55 | 29
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 23 | 11
Application site pruritus (General disorders) | 0 | 1
Asthenia (General disorders) | 3 | 0
Catheter site haematoma (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 1
Catheter site oedema (General disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 4
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 3
Chills (General disorders) | 1 | 1
Cyst (General disorders) | 0 | 1
Discomfort (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 2
Fatigue (General disorders) | 7 | 1
Generalised oedema (General disorders) | 1 | 1
Hyperthermia (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Infusion site erythema (General disorders) | 1 | 3
Infusion site extravasation (General disorders) | 1 | 14
Infusion site oedema (General disorders) | 1 | 0
Infusion site pain (General disorders) | 1 | 5
Infusion site phlebitis (General disorders) | 3 | 4
Infusion site pruritus (General disorders) | 0 | 1
Infusion site rash (General disorders) | 0 | 1
Infusion site reaction (General disorders) | 0 | 1
Infusion site swelling (General disorders) | 1 | 1
Infusion site thrombosis (General disorders) | 0 | 1
Infusion site warmth (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 6 | 2
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 6 | 11
Sensation of foreign body (General disorders) | 1 | 0
Ulcer (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 2
Abscess neck (Infections and infestations) | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial rhinitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Candidiasis (Infections and infestations) | 5 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 2 | 1
Ear infection (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 1 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 4 | 2
Fungal skin infection (Infections and infestations) | 4 | 2
Furuncle (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Genital candidiasis (Infections and infestations) | 2 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Infusion site abscess (Infections and infestations) | 0 | 1
Infusion site cellulitis (Infections and infestations) | 1 | 0
Injection site abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Morganella infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Oral candidiasis (Infections and infestations) | 2 | 2
Oral fungal infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 3
Pelvic abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1
Prostate infection (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 2 | 1
Skin infection (Infections and infestations) | 2 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 2 | 0
Tonsillitis bacterial (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Trichomoniasis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 13 | 7
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 7 | 2
Vulvovaginitis trichomonal (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Wound infection fungal (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 2
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 5 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 4
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood amylase increased (Investigations) | 2 | 2
Blood calcium decreased (Investigations) | 1 | 0
Blood chloride decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 4
Blood culture positive (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 4 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 1 | 1
Blood phosphorus decreased (Investigations) | 0 | 2
Blood potassium decreased (Investigations) | 1 | 1
Blood pressure decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Blood pressure systolic increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 2 | 0
C-reactive protein increased (Investigations) | 1 | 2
Culture wound positive (Investigations) | 0 | 1
Drug level above therapeutic (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 2
International normalised ratio increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Platelet count increased (Investigations) | 3 | 0
Polymerase chain reaction (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 10 | 10
Dysgeusia (Nervous system disorders) | 3 | 1
Essential tremor (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 15 | 19
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 1 | 2
Neurological decompensation (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 2
Post polio syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 5
Tremor (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 5 | 6
Confusional state (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 15 | 16
Restlessness (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 2 | 2
Bladder spasm (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 3
Renal impairment (Renal and urinary disorders) | 3 | 3
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 3
Urine odour abnormal (Renal and urinary disorders) | 1 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 1
Scrotal irritation (Reproductive system and breast disorders) | 0 | 1
Vaginal disorder (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vulval disorder (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 21
Pruritus allergic (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 10 | 9
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 5
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Venipuncture (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 7 | 5
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 3 | 2
Lymphoedema (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Comparing duration of intravenous (IV) therapy for linezolid (LZD) and vancomycin (VAN) in study, participants in LZD group had option to switch to oral therapy while those in VAN group had to remain on IV therapy until completion of study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.